CLINICAL TRIAL: NCT04606589
Title: Feasibility Study Evaluating the Efficacy of a Wireless Vital Signs Monitor for Critically Ill Newborns in Kenya
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Neopenda, PBC (Industry)
Collaborators: Center for Public Health and Development (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MSU/DRPI/MUERC/00864/20
Record Dates: First submitted 2020-10-14; First posted 2020-10-28 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2020-10

CONDITIONS: Newborn Morbidity; Newborn Complication
Keywords: Newborn health; Newborn morbidity; Newborn critical care

STUDY DESIGN:
Intervention Model Description: This is a simple pre/post interventional study model.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard-of-care (No Intervention): The standard-of-care arm will receive intermittent monitoring of pulse rate and blood oxygen saturation with a conventional pulse oximeter. Temperature and respiratory rate will also be monitored intermittently with a digital thermometer and manual counting of breaths respectively.
- neoGuard vital signs monitor (Experimental): The intervention group will receive continuous vital signs monitoring of pulse rate, blood oxygen saturation, temperature and respiratory rate with the neoGuard device.
  Interventions: Device: neoGuard vital signs monitor

INTERVENTIONS:
Device: neoGuard vital signs monitor — The neoGuardTM device is a 4-in-1 wearable vital signs monitor designed to continuously measure temperature, pulse rate, respiratory rate and blood oxygen saturation in newborns.
  Arms: neoGuard vital signs monitor

SUMMARY:
The neoGuard device is a 4-in-1 wearable vital signs monitor designed to continuously measure temperature, pulse rate (PR), respiratory rate (RR) and blood oxygen saturation (SpO2) in newborns. In this study, researchers will evaluate the feasibility of the neoGuard device at two rural health facilities in Western Kenya and assess the preliminary efficacy of the technology in improving health outcomes for newborns.

This is a pre/post intervention study. The standard-of-care arm (n=223) will be enrolled between 20 Oct - 20 Nov, 2020 and the neoGuard intervention arm (n=223) will be enrolled between 1 - 31 Dec, 2020.

ELIGIBILITY:
Inclusion Criteria:

* Age <28 days
* Admitted to the neonatal intensive care unit
* Weight at birth/admission ≥2000 g
* Low-to-moderate disease severity as determined by the Signs of Inflammation in Children that Kill (SICK) score card (SICK score ≤2.4 at admission is eligible)
* Parent/guardian willing to provide informed consent for their newborn to participate in study

Exclusion Criteria:

* Age >28 days
* Has a condition that impairs them from wearing the device, such as hydrocephaly.
* Weight at birth <2000 g
* Very severe disease status (SICK score >2.4 at admission)

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 167 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
In-hospital newborn mortality | From date of admission to date of discharge or referral or death, up to 28 days
  Proportion of deaths that occur during hospital stay.

SECONDARY OUTCOMES:
Complication rate | From date of admission to date of discharge or referral or death, up to 28 days
  Proportion of cases that experience a complication resulting from their underlying illness or a complication resulting from their medical care.
Length of stay in hospital | From date of admission to date of discharge or referral or death, up to 28 days
  Time elapsed between admission and discharge of a patient (measured in days).

OTHER OUTCOMES:
Mean alarm-response time | From date of admission to date of discharge or referral or death, up to 28 days
  Average time elapsed between when each neoGuard alarm goes off and when a nurse attends to the patient (measured in seconds by the Neopenda app).

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Olayo, MD, Principal Investigator — Center for Public Health and Development
Locations (1):
- Kakamega County Referral Hospital, Kakamega, Kenya

IPD SHARING:
Plan to Share IPD: No